CLINICAL TRIAL: NCT03940651
Title: Effect of Spinal Versus General Anesthesia on Cardiac and Renal Biomarker Levels in Hip and Knee Arthroplasty Surgery
Brief Title: Cardiac and Renal Biomarkers in Arthroplasty Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Washington University School of Medicine (Other)
Collaborators: Abbott (Industry); BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201812100
Record Dates: First submitted 2019-04-03; First posted 2019-05-07 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Renal Injury; Anesthesia; Myocardial Injury; Arthropathy of Knee; Arthropathy of Hip
MeSH Terms: interventions — Anesthesia, Spinal; Anesthetics, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Arthroplasty (Experimental): Surgery to replace the knee joint with prothetic joint
  Interventions: Drug: Spinal Anesthesia; Drug: General Anesthetics
- Hip Arthroplasty (Experimental): Surgery to replace the hip joint with prothetic joint
  Interventions: Drug: Spinal Anesthesia; Drug: General Anesthetics

INTERVENTIONS:
Drug: Spinal Anesthesia — Patients will be randomized to type of anesthesia
Drug: General Anesthetics — Patients will be randomized to type of anesthesia

SUMMARY:
The investigators will compare the effect of spinal anesthesia to general anesthesia on the level of high sensitivity cardiac biomarkers in patients undergoing hip or knee arthroplasty. The investigators will also measure renal biomarkers in urine to evaluate kidney injury in the postoperative period.

DETAILED DESCRIPTION:
The study will enroll a total of 140 adult patients undergoing hip or knee arthroplasty (equal numbers) at Barnes-Jewish-Hospital. These procedures will be randomized with 50% of the procedures performed under spinal anesthesia and 50% procedures performed under general anesthesia.

Patients randomized to spinal anesthesia will receive sedation with dexmedetomidine up to 1 mcg/kg/min, and then add small dose of propofol (up to 50 mcg/kg/min) and fentanyl at the discretion of the anesthesia provider the Richmond Agitation and Sedation Scale (RASS) -2 to -3. Headphones to play music will be offered to patients undergoing spinal anesthesia to minimize the noise generated from the surgical intervention.

The investigators will study the effect of spinal anesthesia versus general anesthesia on cardiac biomarker levels in hip and knee arthroplasty population (levels of Hs-cTnI postoperatively compared to baseline values) Also, the incidence of postoperative renal injury using investigational renal biomarkers, Myo-Inositol Oxygenase (MIOX) and Nephrocheck

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 60 years or older
* Ability to provide informed consent
* American Society of Anesthesiologists (ASA) classification II or higher

Exclusion Criteria:

* Hip fracture procedures
* Contraindications to neuraxial anesthesia per The American Society of Regional Anesthesia (ASRA) guidelines
* Procedure anticipated duration is longer than expected planned spinal anesthesia duration

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Incidence of myocardial injury defined by new Hs-cTnI elevation postoperatively | Before discharge (approximately 24 hours after surgery)
  Hs-cTnI increase >50% above the sex-specific 99th percentile upper reference limit
Incidence of myocardial injury defined by new Hs-cTnI elevation postoperatively | at time of postoperative visit (around 2 weeks post discharge)
  Hs-cTnI increase >50% above the sex-specific 99th percentile upper reference limit
Investigate the effect of spinal anesthesia on biomarker levels in hip arthroplasty population | Before discharge (approximately 24 hours after surgery)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Investigate the effect of spinal anesthesia on biomarker levels in hip arthroplasty population | at time of postoperative visit (around 2 weeks post discharge)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Investigate the effect of spinal anesthesia on biomarker levels in knee arthroplasty population | at time of postoperative visit (around 2 weeks post discharge)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Investigate the effect of general anesthesia on biomarker levels in hip arthroplasty population | Before discharge (approximately 24 hours after surgery)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Investigate the effect of general anesthesia on biomarker levels in hip arthroplasty population | at time of postoperative visit (around 2 weeks post discharge)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Investigate the effect of general anesthesia on biomarker levels in knee arthroplasty population | Before discharge (approximately 24 hours after surgery)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Investigate the effect of general anesthesia on biomarker levels in knee arthroplasty population | at time of postoperative visit (around 2 weeks post discharge)
  cardiovascular effect measured by changes in levels of Hs-cTnI postoperatively compared to baseline values
Incidence of postoperative renal injury using investigational renal biomarkers | Before discharge (approximately 24 hours after surgery)
  MIOX, Kidney Injury Molecule-1 (KIM-1), Neutrophil gelatinase-associated lipocalin (NGAL) and Nephrocheck measured in ng/ml
Incidence of postoperative renal injury using investigational renal biomarkers | at time of postoperative visit (around 2 weeks post discharge)
  MIOX, Kidney Injury Molecule-1 (KIM-1), Neutrophil gelatinase-associated lipocalin (NGAL) and Nephrocheck measured in ng/ml

SECONDARY OUTCOMES:
Difference renal biomarkers levels according to anesthesia groups - Pain scores and the incidence of intraoperative hypotension | before discharge
  Pain score assessment using the visual analog score
Difference renal biomarkers levels according to anesthesia groups - Pain scores and the incidence of intraoperative hypotension | at time of postoperative visit (around 2 weeks post discharge)
  Pain score assessment using the visual analog score
Difference renal biomarkers levels according to anesthesia groups - Pain medication consumption and the incidence of intraoperative hypotension | before discharge
  Pain medication consumption measured in mg
Difference renal biomarkers levels according to anesthesia groups - Pain medication consumption and the incidence of intraoperative hypotension | at time of postoperative visit (around 2 weeks post discharge)
  Pain medication consumption measured in mg
Difference in cardiac biomarker levels according to surgical groups - Pain scores, pain medications consumption and the incidence of intraoperative hypotension | before discharge and at time of postoperative visit (around 2 weeks post discharge)
  Pain score assessment using the visual analog score
Difference in cardiac biomarker levels according to surgical groups - Pain scores, pain medications consumption and the incidence of intraoperative hypotension | before discharge
  Pain score assessment using the visual analog score
Difference in cardiac biomarker levels according to surgical groups - Pain scores and the incidence of intraoperative hypotension | at time of postoperative visit (around 2 weeks post discharge)
  Pain score assessment using the visual analog score
Difference in renal biomarker levels according to surgical groups - Pain medication consumption and the incidence of intraoperative hypotension | before discharge
  Pain medication consumption measured in mg
Difference in renal biomarker levels according to surgical groups - Pain medication consumption and the incidence of intraoperative hypotension | at time of postoperative visit (around 2 weeks post discharge)
  Pain medication consumption measured in mg
The effect of nonsteroidal anti-inflammatory drugs (NSAIDs) on renal biomarkers - Pain scores and the incidence of intraoperative hypotension | before discharge
  Pain score assessment using the visual analog score
The effect of nonsteroidal anti-inflammatory drugs (NSAIDs) on renal biomarkers - Pain scores and the incidence of intraoperative hypotension | at time of postoperative visit (around 2 weeks post discharge)
  Pain score assessment using the visual analog score
The effect of nonsteroidal anti-inflammatory drugs (NSAIDs) on renal biomarkers - Pain medication consumption and the incidence of intraoperative hypotension | before discharge
  Pain medication consumption measured in mg
The effect of nonsteroidal anti-inflammatory drugs (NSAIDs) on renal biomarkers - Pain medication consumption and the incidence of intraoperative hypotension | at time of postoperative visit (around 2 weeks post discharge)
  Pain medication consumption measured in mg

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Helwani, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Cram P, Lu X, Kates SL, Singh JA, Li Y, Wolf BR. Total knee arthroplasty volume, utilization, and outcomes among Medicare beneficiaries, 1991-2010. JAMA. 2012 Sep 26;308(12):1227-36. doi: 10.1001/2012.jama.11153. PMID 23011713
- [Background] Khan J, Alonso-Coello P, Devereaux PJ. Myocardial injury after noncardiac surgery. Curr Opin Cardiol. 2014 Jul;29(4):307-11. doi: 10.1097/HCO.0000000000000069. PMID 25029449